CLINICAL TRIAL: NCT03714061
Title: Effects of Pain Neuroscience Education Compared to Self-Management Education for Patients With Chronic Low Back Pain: a Randomized Clinical Trial
Brief Title: Effects of Pain Neuroscience Education vs. Self-Management Education in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Thais Cristina Chaves, Professor PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 66674117.5.0000.5414
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2019-06

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single blind, randomized clinical trial, controlled
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education (PNE) (Experimental): The PNE will be administered following Explaining Pain concepts (Butler and Moseley, 2013), initially contextualizing the importance of the program. The program will be administered as interactive workshops lasting 50 minutes. In addition, the participants were oriented to perform at home a group o motor control exercises during three weeks, twice a week.
  Interventions: Other: Pain Neuroscience Education
- Self-Management Education (SME) (Active Comparator): The SME education will be administered as an interactive workshop lasting 50 minutes. The program is based on the Back-book material (Roland et al, 2011), focusing on concepts targeting change of behavior and beliefs. In addition, the participants were oriented to perform at home a group o motor control exercises during three weeks, twice a week.
  Interventions: Other: Self-Management Education

INTERVENTIONS:
Other: Pain Neuroscience Education — The PNE will be administered following Explaining Pain concepts, initially contextualizing the importance of the program, addressing concepts of neuroscience and pain, incorrect information about what is pain, how the brain responds to nociception in a variety of situations, and how an experience of danger can trigger or aggravate a state of pain, coexistence of several potential protection systems, central sensitization and how to promote behavioral change, abandoning incorrect beliefs, proposing graded activity exposure.
  In addition, participants were requested to perform a group of 7 exercises two times a week. In the day of the education session (second day), participants were again oriented on how to perform the exercises and invited to show the way they were executing them at home. In the first session, participants were trained on how to perform the abdominal bracing and oriented to repeat the maneuver in all exercises during the following three weeks.
  Arms: Pain Neuroscience Education (PNE)
Other: Self-Management Education — Concepts about pain, musculoskeletal pain, chronic pain and disability will be addressed. Participants will be guided on the process of chronic pain, associated suffering, conceptual model of fear-avoidance and clarified on avoidant and confronting profiles. In a third phase, strategies will be presented on how to deal with chronic pain, with advice on the harmful effects of restricting activities and the use of drug therapy in a careful way (Dupeyron et al, 2011).
  In addition, participants were requested to perform a group of 7 exercises two times a week. In the day of the education session (second day), participants were again oriented on how to perform the exercises (reinforcement) and invited to show the way they were executing them at home. In the first session, participants were trained on how to perform the abdominal bracing and oriented to repeat the maneuver in all exercises during the following three weeks.
  Arms: Self-Management Education (SME)

SUMMARY:
Chronic low back pain interventions may include exercises, manual therapy, health education, and pain education, strategies based on psychological or behavioral change approaches, as well as biopsychosocial interventions. Pain self-management programs basically aim to engage the participant in activities, stimulating the patient to be more active in life and live despite the pain. However, pain neuroscience education is a new approach recognized as therapeutic patient education (ETP) and is best described as a form of cognitive rather than behavioral therapy. However, there are few studies in the literature comparing those types pain education. Thus, the purpose of this study will be to compare the immediate effects of an educational program focused on Pain Neuroscience Education vs. Pain self-management educations for patients with chronic low back pain considering the outcomes of pain intensity, catastrophizing and pain self-efficacy.

DETAILED DESCRIPTION:
There is some evidence in the literature suggesting better effects of pain neuroscience than "traditional pain education" based on pain self-management ("living despite the pain") and biomedical models. As the focus is based on cognitive change, pain neuroscience programs could be more effective than pain self-management programs, contributing to reconceptualize beliefs and minimize the level of threatening perceived by the brain. Gallagher et al (2013) reported effects of a pain neuroscience education program based on a book of metaphors compared to a pain self-management program (Back book) and reported greater immediate from pain neuroscience education on pain catastrophizing and pain knowledge. The hypothesis of this study is that a pain neuroscience education will show more effective results for pain intensity, catastrophizing and pain self-efficacy when compared to the pain self-management program in patients with CLBP. The purpose of this study will be to compare the immediate effects of an educational program focused on Pain Neuroscience Education vs. Pain self-management program for patients with chronic low back pain (CLBP) considering the outcomes of pain intensity, catastrophizing and pain self-efficacy. The investigators will recruit 108 with CLBP between 18 and 60 years and both genders. The sample size will be randomized into two arms: fifty participants will be submitted to Pain Neuroscience Education and the remaining fifty to Pain Self-Management education. Both interventions will be administered in one session (50 minutes). The programs will be showed as interactive workshops. Participants will be submitted to a brief initial assessment considering: pain intensity, fear of movement, anxiety and depression, catastrophizing, pain self-efficacy and global perceived effect.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 60 years;
2. Medical diagnosis of nonspecific CLBP in the last 3 months and/or pain at least half of the days in the past 6 months, that is located between T12 and the gluteal folds;
3. Pain intensity equal to or greater than three on numerical pain rating scale (NPRS)
4. Score greater than 14% on the Oswestry Disability Index and
5. Acceptable cognitive function assessed by Mini-Mental examination.

Exclusion Criteria:

1. red flags indicative of systemic involvement;
2. neurological symptoms, psychiatric, rheumatologic and cardiac diseases;
3. active radiculopathy;
4. lumbar stenosis;
5. spondylolisthesis;
6. history of spinal surgeries;
7. pregnancy;
8. previous physical therapy for low back in the past year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity - Numerical Pain Rating Scale (NPRS) | At the beginning of the study (just after the randomization) and 2 weeks after the initial assessment
  The NPRS used to assess pain intensity in this trial will consist in a sequence of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable" (Costa et al, 2008). Previous research has found the NPRS to be responsive to change, with a minimum clinically important difference (MCID) of 2.4 among patients with CLBP receiving exercise or education (Maughan and Lewis, 2010).
Pain catastrophizing - Pain Catastrophizing Scale | At the beginning of the study (just after the randomization) and 2 weeks after the initial assessment
  The PCS translated and validated to Brazilian Portuguese by Sehn et al. (2012) will be used. The scale is composed of 13 items staggered on 6-point ordinal scale (0-5). The total score is the sum of the items divided by the number of items answered, with the minimum score being 0 and the maximum being 5 for each item. Higher scores indicated a greater presence of catastrophizing thoughts. The total score of the scale could vary between 0 and 52 points. A recent systematic review found that catastrophizing to be associated with pain and disability at follow-up in CLBP patients (Wertli et al, 2014).
Pain Self-Efficacy | At the beginning of the study (just after the randomization) and 2 weeks after the initial assessment
  Study participants will be evaluated on self-efficacy related to chronic pain, which can be defined as an individual's confidence he/she can successfully produce desirable results related to living with chronic pain. The PSES has 10 items which are rated on a 7-point ordinal scale (ranging from 0: "not at all confident" to 6: "completely confident"). The maximum score is 60 and higher the score, higher the level of self-confidence of the participant to self-manage their pain. It was adapted and validated to Brazilian Portuguese (Sarda et al, 2007). Previous research showed an effect on self-efficacy using a PNE intervention based on metaphors compared to an intervention using cognitive-behavioral concepts (Gallager et al, 2013).

SECONDARY OUTCOMES:
Low Back Pain Disability - Oswestry Disability Index | At the beginning of the study (just after the randomization) and 2 weeks after the initial assessment
  The Brazilian Portuguese version of Oswestry Disability Index (ODI) (Vigatto et al, 2007) will be used to assess low back pain related disability. This instrument consists of 10 items, each of which has six response options. The total score will be calculated by summing up all the points, with the largest possible sum being 50. Higher the score on the scale, higher the level of pain related disability. This sum will be transformed into a percentage by multiplying it by two. Previous research has found that ODI showed responsiveness to change for patients with CLBP, with MCID of 8 points (Maughan and Lewis, 2010).
Fear avoidance beliefs - The fear avoidance beliefs questionnaire (FABQ) | At the beginning of the study (just after the randomization) and 2 weeks after the initial assessment
  The fear avoidance beliefs questionnaire (FABQ) adapted for Brazilian Portuguese (Abreu et al, 2008) consists of 12 self-response items, rated on a seven-point ordinal scale from 0 (completely disagree) to 6 (completely agree). The construct of the scale is fear-avoidance beliefs related to physical activity and work. The score is obtained for each separate subscale: one that addresses the fears and beliefs of participants related to work or physical activities, respectively. The FABQ-Physical activity ranges from 0 to 24 points and the FABQ-work ranges from 0 to 42 points. Higher the scores, higher the level of fear avoidance beliefs affecting the participant. A recent systematic review (Wertli et al, 2014) showed an association between baseline fear avoidance belief and worst levels of pain and disability in low back pain.
Global Perceived Effect | 2 weeks after the initial assessment
  The global perceived effect (GPE) assesses the self-perception on recovery. In this trial the investigators will use an 11-point scale that ranges from -5 ("vastly worse") through 0 ("no change") to +5 ("completely recovered") and participants are asked: "Compared to when this episode first started, how would you describe your back these days?". A higher score indicates higher perception of recovery from the condition (Costa et al, 2008).
Anxiety and Depression - Hospital Anxiety and Depression Scale | At the beginning of the study (just after the randomization) and 2 weeks after the initial assessment
  HADS (Pais-Ribeiro et al, 2007) will be employed to identify anxiety disorders and depression. HADS was developed to assess symptoms of depression and anxiety. It was translated and validated into Portuguese. The HADS is divided into the anxiety subscale (HADS-A) and the depression subscale (HADS-D), both containing seven interspersed items. It is composed of seven items for depression and seven items for anxiety, each item including four response options ranging from 0 to 3. In this way, the maximum score for depression and anxiety is 21 for each subscale (21 for depression and 21 for anxiety). Each score scale will be considered separately. Higher the scores indicate higher levels of anxiety and depression, however, the cutoff of ≥8 showed good sensitivity and specificity (0.70-0.90) to identify anxiety and depression symptoms compared to the clinical diagnoses (Bjelland et al. 2002).
Exercise Adherence - Exercise Adherence Rating Scale | At the beginning of the study (just after the randomization) and 2 weeks after the initial assessment
  The Exercise Adherence Rating Scale (Beinart et al, 2016) has 10 items which assess adherence to prescribed home exercises. The items are scored using an ordinal scale ranging from totally agree (0) to totally disagree (4), with a maximal score of 64 points. The scale is in process of validation to Brazilian Portuguese. higher overall adherence score indicated better adherence to exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Thais Chaves, PhD, Principal Investigator — Professor - Ribeirão Preto Medical School - University of São Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No